CLINICAL TRIAL: NCT02503397
Title: Latent Iron Deficiency at Birth Influences Auditory Neural Maturation in Late Preterm and Term Infants
Status: Completed | Type: Observational
Sponsor: Sir Ganga Ram Hospital (Other)
Responsible Party: Principal Investigator, Vivek Choudhury, DNB trainee in Neonatology, Sir Ganga Ram Hospital
Other Study IDs: EC/06/10/145
Record Dates: First submitted 2015-07-12; First posted 2015-07-21 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Latent Iron Deficiency at Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Latent iron deficiency: Infants with cord serum ferritin levels ≤ 75 ng/mL
  Interventions: Device: Auditory brainstem evoked response (ABR)
- Normal iron status: Infants with cord serum ferritin levels > 75 ng/mL.
  Interventions: Device: Auditory brainstem evoked response (ABR)

INTERVENTIONS:
Device: Auditory brainstem evoked response (ABR) — Bilateral monaural auditory brainstem response (ABR) test would be recorded in each subject with a Bio-logic Navigator Evoked Response System (Bio-logic Systems, USA) between 24 and 48 hours after birth by an audiologist skilled in administering ABR to newborn infants. ABRs shall be performed using 80 dB nHL broadband click stimuli with insert earphones and with the subject lying supine in a quiet room and normal skin temperature. The clicks would be presented at a repetition rate of 29.9/second, and three runs of 2000 repetitions to be recorded for each ear. The 2 most replicable runs for each ear shall be averaged and used for analysis. Absolute latencies of waves I, III, V and IPL (I-III, III-V, and I-V) shall be measured and considered outcomes

SUMMARY:
This study evaluates auditory neural maturation by auditory brainstem evoked response in late preterm and term infants with in utero iron deficiency compared with neonates with normal in utero iron status.

DETAILED DESCRIPTION:
Iron is an essential nutrient for brain development. During early human development, iron is required for multiple neurodevelopmental processes. To meet the iron requirements of a developing brain, active transfer of iron occurs across the placenta during the last trimester of pregnancy and therefore most term infants have iron replete status at birth. However, maternal iron deficiency during pregnancy, a global health problem, can negatively affect the fetal iron status. In addition, prematurity, maternal diabetes mellitus, preeclampsia, maternal smoking, and intrauterine growth restriction during pregnancy have also been associated with decreased iron transfer to the fetus often leading to in utero iron deficiency.

Cord serum ferritin (SF) level at birth provides a good measurement of fetal tissue iron storage concentration and is therefore often used to evaluate in utero iron status. The absolute and interpeak latencies on auditory brainstem evoked response (ABR) are often used as surrogate outcome measures for neural maturation in the neonates. The absolute latencies for each of these ABR waves and the interpeak latencies (IPL, I-III, III-V, and I-V) are influenced by the degree of myelination, neuronal development, synaptic function, and axonal growth in the auditory nervous system. The absolute latencies and IPL decrease as the auditory neural system matures with age in neonates.

Although iron is essential for auditory neural maturation during the perinatal period, there is a paucity of data regarding the concomitant effect of in utero iron deficiency on auditory neural maturation in late preterm and term infants. The present prospective study is planned with an objective to determine the association of in utero iron deficiency as evaluated by cord ferritin with auditory neural maturation at birth in ≥ 34 weeks GA infants.

ELIGIBILITY:
Inclusion Criteria:

* Neonates born between 34 - 42 weeks of gestation at Sir Ganga Ram Hospital, New Delhi

Exclusion Criteria: Infants with

* craniofacial anomalies
* chromosomal disorders,
* hemolytic disease (coomb's positive),
* multiple gestation,
* history of third trimester maternal infections,
* clinical chorioamnionitis,
* Apgar score < 5 at 5 minutes,
* TORCH infections (toxoplasmosis, other infections, rubella, cytomegalovirus infection and herpes simplex),
* clinical or culture proven sepsis,
* admission to the Neonatal Intensive Care Unit,
* infants on whom cord blood not collected and on whom ABR could not be performed

Ages: 1 Day to 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All neonates born between 34 - 42 weeks of gestation at Sir Ganga Ram Hospital during study period would be evaluated for enrolment in the study till 30 neonates each enrolled in the three groups: appropiate for gestational age, small for gestational age, infants of diabetic mother.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2011-07; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Auditory neural maturation | 3 days
  Auditory neural maturation as assessed by auditory brainstem response at birth in≥ 34 weeks gestational age infants with normal in utero iron status compared with infants with in utero latent iron deficiency

REFERENCES:
- [Derived] Choudhury V, Amin SB, Agarwal A, Srivastava LM, Soni A, Saluja S. Latent iron deficiency at birth influences auditory neural maturation in late preterm and term infants. Am J Clin Nutr. 2015 Nov;102(5):1030-4. doi: 10.3945/ajcn.115.113084. Epub 2015 Aug 26. PMID 26310540